CLINICAL TRIAL: NCT02047955
Title: Tornier Shoulder Outcomes Clinical Study
Brief Title: Tornier Shoulder Outcomes Study to Examine Safety and Functional Outcomes in Shoulder Arthroplasty and Fracture Patients
Status: Terminated | Type: Observational
Why Stopped: Sponsor business decision
Sponsor: Stryker Trauma and Extremities (Industry)
Responsible Party: Sponsor
Other Study IDs: 13B-T-SHOULDER-RM
Record Dates: First submitted 2014-01-24; First posted 2014-01-29 (Estimated); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Shoulder Arthroplasty and Fracture Repair
MeSH Terms: interventions — Arthroplasty, Replacement, Shoulder; Fracture Fixation, Internal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Shoulder Arthroplasty — Data will be collected for commercially available Sponsor devices. These systems treat both the humeral and glenoid side of the shoulder joint. The following products will be included in the study in the geographies where they are commercially available.
  * Aequalis Ascend Flex Convertible Shoulder System
  * Pyrocarbon Humeral Head (used with Aequalis Ascend Flex)
  * Simpliciti Shoulder Prosthesis
  * Aequalis Reversed Fracture Prosthesis
  * Aequalis PerFORM Glenoid
  * Aequalis PerFORM+ Glenoid
  * Aequalis PerFORM Reversed Glenoid
  Devices previously included, but discontinued under clinical investigation plan (CIP) version 4.0:
  * Aequalis Resurfacing Head
  * Aequalis Ascend Anatomic Shoulder System
  * Aequalis IM Humeral Nail - Short and Long
  * ORTHOLOC™ SPS (Shoulder Plating System)
  * Aequalis Reversed II Shoulder System
  * Aequalis Adjustable Reversed Prosthesis
  * Aequalis Flex Revive Shoulder System
  Other Names: Osteosynthesis

SUMMARY:
The Tornier Shoulder Outcomes Study is designed to collect safety and efficacy data on designated commercially available Tornier Shoulder repair products. In addition, this study will provide performance data for use in education, marketing materials, peer-reviewed publications and support research and development of future products.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Willing and able to comply with the requirements of the study protocol
* Considered for treatment with one or more Tornier shoulder arthroplasty or fracture devices included in this study

Exclusion Criteria:

* Patients who are not able to comply with the study procedures based on the judgment of the assessor will be excluded (e.g. cannot comprehend study questions, inability to keep scheduled assessment times)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from United States and Europe
Sampling Method: Non-Probability Sample
Enrollment: 7500 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2024-09-12 (Actual); Study Completion 2024-10-16 (Actual)

PRIMARY OUTCOMES:
Number of device associated and procedure associated adverse events | up to 10 years
  Adverse events will be evaluated from inclusion to last follow-up and will be documented during the study and categorized as whether they are serious and whether they are related to the Sponsor device or implant procedure.

SECONDARY OUTCOMES:
Rates of reoperation and revision surgery | up to 10 years
  The cumulative incidence of device revisions and reoperations will be reported as well as Kaplan-Meier estimates for implant survival at the end of the clinical investigation.

OTHER OUTCOMES:
Time to first revision surgery | up to 10 years
  Time from primary study surgery to revision surgery
Change from baseline and previous visit in ASES scores | at 1, 2, 5, 7, and 10 years of follow-up
  ASES Score = American Shoulder and Elbow Surgeons Score
Constant Score | at 1, 2, 5, 7, and 10 years of follow-up
  The total score by visit and the within subject score changes of the Constant Total Score from visit to visit will be analyzed to help identify the changes on the subject level. This analysis will be part of the final report.
Change from baseline and previous visit in SANE scores | at 1, 2, 5, 7, 10, 15, and 20 years follow-up
  SANE = Single Assessment Numeric Evaluation
Subject Satisfaction | at 1, 2, 5, 7, and 10 years of follow-up
  The total score by visit and the within subject score changes of the Patient Satisfaction Score from visit to visit will be analyzed to help identify the changes on the subject level (assessed as improved, worsened or no change). This analysis will be part of the final report.
Cumulative incidence of migration, radiolucency, osteolysis, and bone wear | at 1, 2, 5, 7, and 10 years of follow-up
  as assessed by available X-ray, CT, or MRI
EQ-5D-5L | at 1, 2, 5, 7, and 10 years of follow-up
  The total score by visit and the within subject score changes of the EQ-5D-5L from visit to visit will be analyzed to help identify the changes on the subject level (assessed as improved, worsened or no change). This analysis will be part of the final report.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Gibson, Study Director — Stryker Trauma & Extremities
Locations (15):
- United States (15):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - California Pacific Orthopaedics, San Francisco, California
  - Western Orthopaedics, Denver, Colorado
  - Resurgens Orthopaedics, Atlanta, Georgia
  - University of Iowa Sports Medicine Clinic, Iowa City, Iowa
  - Lexington Clinic Orthopedics - Sports Medicine Center, Lexington, Kentucky
  - Great Lakes Orthopaedic Center, Traverse City, Michigan
  - Allina Health Orthopedics, Edina, Minnesota
  - University of MO - Columbia, Columbia, Missouri
  - Jersey Medical Center, Jersey City, New Jersey
  - Duke University, Durham, North Carolina
  - Rothman Institute Orthopaedics, Philadelphia, Pennsylvania
  - Ascension Medical Group Seton Orthopedics, Austin, Texas
  - UT Southwestern, Dallas, Texas
  - Fondren Orthopedic Group, Houston, Texas

IPD SHARING:
Plan to Share IPD: No